CLINICAL TRIAL: NCT07324486
Title: Comparison of Functional Outcomes and Postoperative Analgesic Efficacy Between Adductor Canal Block + IPACK Block and Adductor Canal Block + Genicular Nerve Block in Patients Undergoing Total Knee Arthroplasty
Brief Title: Postoperative Analgesic Efficacy Between Adductor Canal Block + IPACK Block and Adductor Canal Block + Genicular Nerve Block in Total Knee Arthroplasty
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Konya Beyhekim Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Sami Uyar, Dr., Konya Beyhekim Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KonyaBeyhekimTRH2025/0115
Record Dates: First submitted 2025-12-10; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Total Knee Arthroplasty; Adductor Canal Block; Genicular Nerves Block; IPACK Block Multimodal Analgesia
Keywords: total knee arthroplasty; adductor canal block; genicular nerves block; IPACK

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: single blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP IPACK (Other): ADDUCTOR CANAL BLOCK + IPACK
  Interventions: Drug: Adductor Canal Block (ACB) + iPACK Block
- GROUP GENİCULAR (Experimental): ADDUCTOR CANAL BLOCK + GENİCULAR BLOCK
  Interventions: Drug: adductor canal block + genicular blocks

INTERVENTIONS:
Drug: Adductor Canal Block (ACB) + iPACK Block — Patients who underwent total knee arthroplasty surgery with IPACK + adductor canal block , 25 patients. After the needle tip is placed in the target area between the popliteal artery and the femur, the local anesthetic solution (10 ml of 0.5% bupivacaine + 10 ml of physiological saline) is slowly injected after negative aspiration. After the needle tip is placed within the adductor canal, the local anesthetic solution (10 ml of 0.5% bupivacaine + 10 ml of physiological saline) is slowly injected after negative aspiration.
  Arms: GROUP IPACK
Drug: adductor canal block + genicular blocks — Patients who underwent total knee arthroplasty surgery with genicular blocks + adductor canal block , 25 patients. The tip of the needle is directed toward the superior lateral, superior medial, and inferior medial genicular nerves under ultrasound guidance.2 ml of local anesthetic (0.5% bupivacaine) is injected into each nerve region. After the needle tip is placed into the adductor canal, the local anesthetic solution (10 ml of 0.5% bupivacaine + 10 ml of physiological saline) is slowly injected after negative aspiration.
  Arms: GROUP GENİCULAR

SUMMARY:
The aim of this study is to compare the postoperative analgesic efficacy and functional outcomes of the IPACK+Adductor Canal Block with the Genicular Nerve Block+Adductor Canal Block block in patients undergoing total knee arthroplasty (TKA). The primary objective (measurable) is to evaluate functional improvement using 6-Clicks scores, while secondary objectives include pain scores (Vas Score), opioid consumption, hospital stay duration, and patient satisfaction (Patient Satisfaction Index).

IPACK : The infiltration between the popliteal artery and capsule of the knee

DETAILED DESCRIPTION:
Group I: Patients who underwent IPACK + Adductor canal block after TDA surgery Group G: Patients who underwent Genicular nerve block + Adductor canal block after TDA surgery

This study will be designed as a prospective randomized trial, and randomization will be performed using the sealed envelope method. This method will be carried out as follows:

First, the study will include two groups: Group I (patients who received a block between the posterior knee capsule and the popliteal artery (IPACK) + adductor canal block (AKB)) and Group G (patients who received a genicular nerve block + adductor canal block). The number of subjects in each group will be adjusted to be equal.

Simple randomization: A list will be created to assign subjects to groups using software (e.g., the RANDBETWEEN function in Excel or an online randomization tool) or a random number table. Each participant will be assigned a serial number in the randomization list (e.g., from 1 to 100). Group Assignment: A group assignment is determined for each number in the randomization list. A random sequence number will be written on each envelope. A piece of paper containing the group assignment corresponding to the number will be placed inside the envelope (e.g., "Group I" or "Group G").

The envelopes will be securely sealed and sealed to prevent any crossover between groups. The prepared envelopes will be randomly mixed.

When each participant is included in the study, an envelope will be opened in sequence.

The participant will be assigned to the relevant group according to the information in the envelope. Since the study requires blinding, no one other than the person opening the envelope will know the group assignment. The envelopes will be prepared by a person not involved in the study.

They will be divided into Group I (IPACK+AKB) and Group G (GENIKÜLER+AKB); additionally, clinicians performing IPACK+AKB and Geniküler+AKB will not be involved in the postoperative data collection period. This research study will be limited to TDA surgeries. ASA 1-2-3 TDA surgeries performed in orthopedic operating rooms will be included.

Study Design According to randomization, all patients will undergo a standard spinal anesthesia protocol administered by anesthesiologists with at least 5 years of clinical experience who are blinded to the randomization.

This study will be designed as a prospective randomized study, and randomization will be performed using a sealed envelope method.

Patients will be divided into Group I (IPACK+AKB) and Group G (Genicular+AKB); additionally, clinicians performing IPACK+AKB and Genicular +AKB will not be included in the postoperative data collection period. This research study will be limited to TDA surgeries. ASA 1-2-3 risk patients will be included.

Standard monitoring procedures will be performed on all patients, including electrocardiography (ECG), peripheral oxygen saturation (SpO2), and noninvasive arterial blood pressure monitoring. Patients will be monitored according to ASA-defined criteria, and after vital signs are observed, the anesthesiologist will administer 1 mg of midazolam intravenously for sedation, followed by spinal anesthesia using a 25-gauge spinal needle and 12.5 mg of bupivacaine. Depending on randomization, the block will be performed according to the group after the surgery is completed. Information about the operation and the patient will be recorded perioperatively.

After postoperative monitoring, the patient will be positioned, and then, according to randomization, IPACK+AKB or Genicular+AKB will be performed with ultrasound guidance. For Group I, the linear probe will be placed with the patient in the supine position and the knee slightly flexed. The linear probe is placed in the transverse plane in the upper part of the popliteal region, where the popliteal artery is visible. The femoral condyles, popliteal artery, and target injection site (the space between the popliteal artery and the femur) are visualized with ultrasound. After ensuring sterile conditions, the needle is advanced laterally to medially, parallel to the ultrasound probe. After the needle tip is placed in the target area between the popliteal artery and the femur, the local anesthetic solution (10 ml of 0.5% bupivacaine + 10 ml of physiological saline) is slowly injected after negative aspiration. After completing the IPACK Block, a high-frequency linear probe is placed in the transverse plane in the middle of the thigh, in the area where the femoral artery can be palpated. The sartorius muscle, femoral artery, and structures within the adductor canal (such as the saphenous nerve) are identified on the ultrasound image. After ensuring sterile conditions, the needle is advanced laterally to medially, parallel to the ultrasound probe. After the needle tip is placed within the adductor canal, the local anesthetic solution (10 ml of 0.5% bupivacaine + 10 ml of physiological saline) is slowly injected after negative aspiration. This completes the AKB.

Patients in Group G are positioned supine with the knee slightly bent. The injection site is cleaned with an antiseptic solution and a sterile field is established. A high-frequency linear ultrasound probe is placed over the medial and lateral regions of the knee joint. The condyles of the femur and tibia, arteries, and areas where the genicular nerves pass are identified on the ultrasound image. Under sterile conditions, the block needle is advanced subcutaneously parallel to the ultrasound probe (in-plane technique). The tip of the needle is directed toward the superior lateral, superior medial, and inferior medial genicular nerves under ultrasound guidance. When the needle tip reaches the vicinity of the targeted nerve, negative aspiration is performed to ensure that it is not within a vessel. Subsequently, 2 ml of local anesthetic (0.5% bupivacaine) is injected into each nerve region. After all injections are completed, the needle is removed, and a sterile bandage is applied to the injection sites. After the genicular nerve block is completed, a high-frequency linear probe is placed in the transverse plane in the middle of the thigh, in the area where the femoral artery can be palpated. The sartorius muscle, femoral artery, and structures within the adductor canal (such as the saphenous nerve) are identified on the ultrasound image. After ensuring sterile conditions, the needle is advanced laterally to medially, parallel to the ultrasound probe. After the needle tip is placed into the adductor canal, the local anesthetic solution (10 ml of 0.5% bupivacaine + 10 ml of physiological saline) is slowly injected after negative aspiration. This completes the AKB.

The VAS score will be recorded in the postoperative recovery room at 30 minutes. After postoperative follow-up, patients will be sent to the ward. All patients in the ward will undergo VAS assessment (at 6, 12, 24, 36, 48, 60, and 72 hours), and intravenous paracetamol 15 mg/kg and intravenous diclofenac 1.5 mg/kg (maximum 75 mg) every 12 hours will be administered. If the VAS score is 4 or higher in the postoperative period, intravenous tramadol 1 mg/kg will be administered as rescue analgesia. This analgesia protocol is routinely applied by the Orthopedics clinic after total knee replacement surgeries; no additional analgesics specific to the study will be administered.

The primary outcome measure of the study is the 6-Clicks score, while the secondary outcome measures are the visual analog scale (VAS) score, total opioid consumption, patient satisfaction (Patient Satisfaction Index), and length of hospital stay.

The 6-Clicks score will be assessed at 6, 12, 24, 36, 48, 60, and 72 hours. The Visual Analog Scale (VAS) score will be recorded at 30 minutes in the postoperative recovery room and at 6, 12, 24, 36, 48, 60, and 72 hours. In addition, total opioid consumption in the first 24 hours, patient satisfaction (Patient Satisfaction Index), and length of hospital stay will also be recorded.

Demographic data (age, height, gender, weight), ASA physical score, and duration of surgery are other data that will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for spinal anesthesia with TDA.
2. Age ≥18.
3. American Society of Anesthesiologists (ASA) physical status score I-III.
4. Patients capable of providing informed consent.

Exclusion Criteria:

1. Active infection at the injection site.
2. Coagulopathy or systemic sepsis.
3. Severe hypovolemia.
4. Patients who refuse regional anesthesia.
5. Known allergy to local anesthetics.
6. Cognitive impairment or uncooperative patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
6-Clicks score | 6.,12.,24.,36.,48.,60.,72. hours
  Known as "6-Clicks" due to being composed of six scored patient activity questions, a patient's "6-Clicks" score falls on a 6- to 24-point scale where a score of 6 represents total functional impairment and a score of 24 represents total absence of impairment.

SECONDARY OUTCOMES:
visual analog scale | Postoperative recovery room 30 minutes and at 6., 12., 24., 36., 48., 60., and 72. hours
  The Visual Analogue Scale (VAS) is a psychometric instrument used in research and clinical studies to measure the intensity of subjective experiences that cannot be objectively quantified using defined biomarkers, such as pain, fatigue, or mood. It typically consists of a 100 mm straight line with descriptive anchors at each end representing the extremes of the sensation (for example, "no pain" at one end and "the most severe pain imaginable" at the other).
total opioid consumption | total opioid consumption 24.hour
  total opioid consumption per day
The Patient Satisfaction Index | first 24. hour
  The Patient Satisfaction Index (PSI) was used to describe self-evaluation of the outcome and responseof 1 or 2 was considered to indicate a satisfying outcomeand 3 or 4 to indicate a dissatisfied outcome.

IPD SHARING:
Plan to Share IPD: No